CLINICAL TRIAL: NCT06103617
Title: Safety and Superiority of Penicillamine in Radiosensitization of Recurrent Head and Neck Cancer: a Single-center, Single-arm, Phase II Clinical Trial
Brief Title: Safety and Superiority of Penicillamine in Radiosensitization of Recurrent Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-416
Record Dates: First submitted 2023-10-15; First posted 2023-10-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer; Recurrent Cancer
Keywords: radiotherapy; radiosensitizer; penicillamine; copper
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — Penicillamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penicillamine group (Experimental): Participants in this group are treated with Penicillamine (250mg each time, 4 times per day) during reradiation.
  Interventions: Drug: Penicillamine

INTERVENTIONS:
Drug: Penicillamine — Participants in this group are treated with Penicillamine (250mg each time, 4 times per day) during reradiation.

SUMMARY:
Our preclinical study confirmed that copper accumulation can lead to radioresistance in vitro and in vivo, and reducing the concentration of copper with copper chelator help to overcome radioresistance. Therefore, the investigators plan to carry out a prospective interventional phase II clinical trial to explore the safety and efficacy of penicillamine (a common copper chelator) as a radiosensitizer in the treatment of recurrent head and neck cancer.

DETAILED DESCRIPTION:
Head and neck cancer is the sixth most common cancer worldwide. Radiotherapy is an important measure to control tumor recurrence. Although radiotherapy has been widely used in patients with head and neck cancer, the 2-year local recurrence rate of patients with locally advanced disease is still as high as 50%-60%. This is associated with a lower radiosensitivity in head and neck cancer. High doses of reirradiation (>60 Gy) are associated with severe late complications and treatment-related mortality. Therefore, finding an appropriate sensitizer to improve the radiosensitivity is the key to improve the survival of recurrent patients. Our preclinical study confirmed that copper accumulation can lead to radioresistance in vitro and in vivo, and the results were published in J Hepatol (IF=25.7). Penicillamine is a commonly used copper chelator in clinical practice and can reduce the concentration of copper in the body. Based on this, the investigators plan to carry out a prospective interventional phase II clinical trial to explore the safety and efficacy of penicillamine as a radiosensitizer in the treatment of recurrent head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent
2. The age is 18-75 years
3. Previously received standard radical radiotherapy or chemoradiotherapy
4. Head and neck tumors with in situ or cervical lymph node recurrence confirmed by pathological biopsy and imaging examination
5. ECOG PS：0/1
6. Laboratory examination confirmed good organ function, which should be carried out within 10 days before the first treatment.

Exclusion Criteria:

1. After evaluation, it does not meet the indications of re-radiotherapy
2. Unable to take oral medication
3. Pregnancy or lactation
4. Known allergy to penicillamine
5. Patients who are judged by the researcher as unsuitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 month
  The objective response rate (ORR) is the proportion of patients who achieve a prespecified reduction in tumor volume that is maintained for a minimum duration. The objective response rate was defined as the sum of complete response plus partial response (CR+PR). According to RECIST1.1 criteria, CR was defined as the disappearance of target lesions and the reduction of the short diameter of pathological lymph nodes to less than 10mm. PR: the sum of the measured diameters of the target lesions reduced by 30% compared with the baseline; PD: the sum of the major diameters of all target lesions increased by at least 20%, and the absolute value of the sum of the major diameters increased by more than 5mm, or new lesions appeared. SD: Changes between PR and PD.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  OS was defined as the time from the date of inclusion until death from any cause.
local-relapse free survival (LRFS) | 2 years
  LRFS was defined as the time from the date of inclusion until tumor relapse.
Incidence of Treatment-Emergent Adverse Events | During treatment and 12 weeks after penicillamine treatment
  treatment-related adverse events will be assessed by CTCAE v5.0

OTHER OUTCOMES:
the biomarkers correlated with ORR, LRFS and OS | 2 years
  The correlations between ORR, OS, LRFS and PD-L1 expression in tissues, tumor mutation burden, tumor-related gene changes, plasma cytokines or other biomarkers were explored.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, M.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - Southern medical university, Guangzhou, Guangdong
  - Nanfang Hospital, Sourthern Medical University, Guangzhou